CLINICAL TRIAL: NCT03402438
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of a Single Oral 25 mg BAY 1142524 IR Tablet Dose in Male and Female Subjects With Renal Impairment and in Age-, Gender-, and Weight-matched Healthy Subjects in a Single Center, Non-controlled, Open-label, Observational Design
Brief Title: Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18106; 2017-003301-17 (EudraCT Number)
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Clinical Trial, Phase I
MeSH Terms: interventions — fulacimstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal (healthy subjects) (Experimental): Healthy subjects matched for age, body weight and gender to the groups with renal impairment
  Interventions: Drug: Fulacimstat (BAY1142524)
- Mildly renal impaired (Experimental): Subjects with renal impairment and an estimated glomerular function rate between equal or above 60 and below 90 ml/min/1.75 m*2
  Interventions: Drug: Fulacimstat (BAY1142524)
- Moderately renal impaired (Experimental): Subjects with renal impairment and an estimated glomerular function rate between equal or above 30 and below 60 ml/min/1.75 m*2
  Interventions: Drug: Fulacimstat (BAY1142524)
- Severely renal impaired (Experimental): Subjects with renal impairment and an estimated glomerular function rate between below 30 ml/min/1.75 m*2
  Interventions: Drug: Fulacimstat (BAY1142524)

INTERVENTIONS:
Drug: Fulacimstat (BAY1142524) — single oral dose of 25 mg immediate-release tablet BAY1142524

SUMMARY:
The study will investigate the pharmacokinetics of BAY1142524 in subjects with mild to severe renal impairment compared to age; weight, and gender-matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 18 to 34 kg/m² (both inclusive)
* Men or confirmed postmenopausal women (by medical report verification and defined as exhibiting natural amenorrhea for at least 12 months before screening or as exhibiting natural amenorrhea for at least 6 months before screening with documented serum follicle-stimulating hormone levels >40 mIU/mL, provided that no prior hormonal treatment has taken place) or women without childbearing potential based on surgical treatment at least 6 weeks before screening such as bilateral tubal ligation, bilateral oophorectomy or hysterectomy (documented by medical report verification).
* Subjects with renal impairment:

eGFR <90 mL/min/1.73 m*2 determined from serum creatinine 2 -10 days prior to dosing.

Stable renal disease, i.e. a serum creatinine value determined at least 3 months before the pre-study visit (e.g. during routine diagnostics) should not vary by more than 20% from the serum creatinine value determined at the pre-study visit

- Healthy subjects eGFR ≥90 mL/min/1.73 m*2 determined from serum creatinine 2 -10 days prior to dosing.

Needs to be within the required age and body weight range of Group 1 (which should not vary by more than+- 10 years and +-10 kg to Groups 2-4).

Exclusion Criteria:

* Clinically relevant findings(e.g. blood pressure, electrocardiogram, ECG; physical examination,laboratory examination)
* Relevant impairment in liver function.
* Pre-existing diseases (including impairment of liver function) for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Any organ transplant < 1 year before participation in this study.
* Subject under dialysis or planned to start dialysis during participation in the study.
* Failure of any other major organ system other than the kidney.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity after single (first) dose (AUC) of BAY1142524 | Pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,6,8,10,12,15,24,36,48,96hours post dose
  AUC(0-tlast) will be used if mean AUC(tlast ∞) >20% of AUC)
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of BAY1142524 | Pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,6,8,10,12,15,24,36,48,96hours post dose
AUC of unbound drug (AUCu) of BAY1142524 | Pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,6,8,10,12,15,24,36,48,96hours post dose
  AUC (0-tlast) u will be used if mean AUC (tlast ∞) >20% of AUC). An additional blood sample for fu will be collected at 2 hours after dosing.
Cmax of unbound drug (Cmax,u) of BAY1142524 | Pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,6,8,10,12,15,24,36,48,96hours post dose
  An additional blood sample for fu will be collected at 2 hours after dosing.

SECONDARY OUTCOMES:
Number of subject with treatment emergent adverse events (TEAEs) as a measure of safety and tolerability | up to 10 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/